CLINICAL TRIAL: NCT07077356
Title: Application of mRNA Vaccine in Liver Transplantation for Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Jiyan Liu, Deputy Director of the Department of Tumor Biological Therapy, West China Hospital, Sichuan University, West China Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HBV mRNA-Liver Tx
Record Dates: First submitted 2025-07-13; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Hepatocellular Carcinoma; Liver Transplantation
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HBV mRNA vaccine, Dose 1 (Experimental)
  Interventions: Biological: HBV mRNA vaccine
- HBV mRNA vaccine, Dose 2 (Experimental)
  Interventions: Biological: HBV mRNA vaccine
- HBV mRNA vaccine, Dose 3 (Experimental)
  Interventions: Biological: HBV mRNA vaccine
- HBV mRNA vaccine, Dose 4 (Experimental)
  Interventions: Biological: HBV mRNA vaccine

INTERVENTIONS:
Biological: HBV mRNA vaccine — HBV mRNA vaccine

SUMMARY:
The therapeutic options for HCC include hepatectomy, liver transplantation, local ablation therapy, transarterial chemoembolization (TACE), radiotherapy, and systemic therapy. However, as early-stage HCC often presents with no obvious symptoms or atypical clinical manifestations, over 80% of patients are diagnosed at an advanced stage, losing the opportunity for surgical resection and leaving liver transplantation as the only potentially curative option. Nevertheless, even after liver transplantation, the recurrence rate of HCC remains as high as 30-45%. In recent years, with the successive launch of novel targeted drugs and immune checkpoint inhibitors, Chinese patients with HCC have gained more treatment options for both disease management and recurrence prevention. However, given the heterogeneity of HCC, only a subset of patients benefit from these therapies.

Hepatitis B virus (HBV) infection is the primary risk factor for HCC, accounting for at least 50% of global HCC cases. In regions with high HBV prevalence-such as East and Southeast Asia, as well as sub-Saharan Africa-the proportion is even higher. While HBV-related HCC can be prevented through vaccination against HBV infection, no specific precision therapy currently exists for patients already diagnosed with HBV-positive HCC. Given that nucleic acid vaccine technology demonstrates value not only in disease prevention but also in immunotherapy-particularly mRNA therapeutic vaccines-this approach holds promise.

mRNA therapeutic vaccines represent a highly promising new modality for tumor treatment. They offer advantages such as excellent safety, long-term expression, and sustained antigen presentation. Additionally, they can mimic the natural infection process of viruses to activate the immune system, eliciting robust immune responses against tumors. Currently, no mRNA therapeutic vaccines targeting HBV-related antigens have been approved for marketing. This HBV mRNA injection is an mRNA therapeutic vaccine encoding HBV-related specific antigens. Its active ingredient consists of modified mRNA encoding HBV-related antigen proteins, formulated into an injectable preparation via lipid nanoparticle (LNP) encapsulation. Preclinical safety evaluations have demonstrated that this vaccine exhibits low toxicity and good tolerability. Building on these preliminary results, this study aims to further evaluate its potential.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥18 years;
* Patients with histologically, cytologically, or clinically diagnosed hepatocellular carcinoma (HCC);
* Patients who, based on the investigator's assessment, meet the indications for liver transplantation and have expressed willingness to undergo transplantation, with a need for bridge therapy or downstaging therapy during the transplant waiting period as evaluated by the investigator;
* Positive for hepatitis B surface antigen (HBsAg) in peripheral blood;
* Eastern Cooperative Oncology Group (ECOG) performance status score: 0-2; (Additional inclusion criteria may be supplemented.)

Exclusion Criteria:

* History of other malignancies, except for adequately treated and non-recurrent within 5 years prior to screening basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, cervical carcinoma in situ, or gastrointestinal mucosal carcinoma, which the investigator deems eligible for inclusion;
* History of or current hepatic encephalopathy; known central nervous system (CNS) metastases that are untreated or not effectively controlled by prior therapy;
* Clinically significant ascites requiring therapeutic intervention at present;
* Known clinically significant uncontrolled cardiac symptoms or diseases;
* Any active autoimmune disease or history of autoimmune diseases, including but not limited to: neurologic diseases related to immunity, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barré syndrome, myasthenia gravis, systemic lupus erythematosus (SLE), connective tissue disorders, scleroderma, inflammatory bowel disease (including Crohn's disease and ulcerative colitis), autoimmune hepatitis, toxic epidermal necrolysis (TEN), or Stevens-Johnson syndrome (excluding type 1 diabetes mellitus controlled with stable-dose insulin); (Additional exclusion criteria may be supplemented.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) and their incidence rates | During one year after initial treatment
Safety: Type, frequency, and severity of treatment-related adverse events as assessed by CTCAE V5.0 | During one year after initial treatment

SECONDARY OUTCOMES:
Objective response rate (ORR) | During one year after initial treatment
Disease control rate (DCR) | During one year after initial treatment
1-year survival rate | During one year after initial treatment
Immunogenicity: The level of antigen-specific T cells | During one year after initial treatment

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, China

IPD SHARING:
Plan to Share IPD: Undecided